CLINICAL TRIAL: NCT00375232
Title: Effects of Montelukast on Occult Exercise-Induced Bronchospasm in Athletes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: EMOEBA Trial
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Exercise-Induced Bronchospasm
Keywords: Exercise-Induced Bronchospasm; Asthma; Cardiopulmonary Stress Test; Eucapnic Voluntary Hyperventilation; Induced sputum
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma

INTERVENTIONS:
Drug: Administration of montelukast or placebo

SUMMARY:
The purpose of this study is to determine if treatment of exercise-induced Bronchospasm with montelukast will help college athletes train more effectively and thus become more competitive in a non ergogenic manner.

DETAILED DESCRIPTION:
Exercise-Induced Bronchospasm (EIB) affects between 7-30% of highly trained athletes. The first phase of this study is to screen varsity level college athletes for EIB using Eucapnic hyperventilation (EVH). Those athletes who screen positive, will be enrolled in phase two, a randomized double-blinded placebo controlled double crossover study. At enrollment, athletes will undergo a cardiopulmonary stress test (CPST) and induced sputum sampling and will then be prescribed daily montelukast/placebo for a three week period. Athletes will return after three weeks and repeat the EVH, CPST, and induced sputum. They will then have a one week washout period followed by crossover once again to daily montelukast/placebo for another three weeks. After the second three weeks they will once again return for a final EVH, CPST, and induced sputum. The goal of this study is to demonstrate that effectively blunting the EIB response with montelukast, indices of ventilation,exercise tolerance, and perhaps overall physical fitness improve, allowing athletes to train more effectively, in a nonergogenic manner.

ELIGIBILITY:
Inclusion Criteria:

* College level varsity athlete
* age 18yr or older
* healthy.
* Able to swallow pills
* No prior history of asthma

Exclusion Criteria:

* Younger than 18yr
* smoker
* Prior history of asthma
* Unable to swallow pills

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Effective blunting of the EIB response by Spirometric measurement
Improvement in indices of ventilation and cardiopulmonary response measured on CPST

CONTACTS AND LOCATIONS:
Overall Officials: Mark O Farber, M.D., Principal Investigator — Indiana University School of Medicine Division of Pulmonary Critical Care and Occupational medicine
Locations (1):
- National Institue Of Fitness and Sport, Indianapolis, Indiana, United States